CLINICAL TRIAL: NCT06505304
Title: Endoscopic Multimodal Assessment Using Advanced Imaging Integrated AI to Predict Recurrence in pOSt-oPerativE CRohn's Disease - PROSPER Study
Brief Title: AI-enabled Endoscopic Prediction of Post-operative Recurrence in Crohn's Disease
Acronym: PROSPER
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: APC188
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; Artificial Intelligence; Virtual Chromoendoscopy; Confocal laser endomicroscopy; OMIC; Machine Learning; Post-operative recurrence
MeSH Terms: conditions — Crohn Disease | interventions — Colonoscopy; Defecation; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intestinal biopsies, Blood, Stool, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-operative CD: Patients undergoing surgery or with a previous (within 3 months from the enrolment) surgery for CD
  Interventions: Procedure: Colonoscopy; Procedure: Intestinal biopsies; Procedure: Confocal laser endomicroscopy; Procedure: Intestinal ultrasound; Diagnostic Test: Stool; Diagnostic Test: Blood; Diagnostic Test: Saliva; Other: Clinical follow-up

INTERVENTIONS:
Procedure: Colonoscopy — The colonoscopy will be performed at 3 or 6 months after surgery according to FC:
  * In patients with FCP >=150µg/g at around 3 months after surgery, a colonoscopy will be immediately performed
  * In patients with FCP <150µg/g at around 3 months after surgery, the colonoscopy will be organized at 6 months after surgery
  Colonoscopy will be performed using high definition white-light endoscopy (HD-WLE) followed by virtual chromoendoscopy (VCE). The neoterminal ileum, ileocolic anastomosis and right colon will be assessed.
  A follow-up colonoscopy will be performed within 18 months after index colonoscopy, as standard of care.
Procedure: Intestinal biopsies — During index colonoscopy, at least 2 biopsies from each of the segments will be taken as standard of practice to assess inflammation in post-operative CD. Only in Irish sites, twelve biopsies - four in the area of ileocolonic anastomosis, four in the neo-terminal ileum and four in the colon just distal to the anastomosis- will be taken for research purposes, in addition to standard-of-care biopsies.
Procedure: Confocal laser endomicroscopy — pCLE with fluorescein injection will be performed during index colonoscopy, in centres where is available, to assess early alteration of the barrier function.
Procedure: Intestinal ultrasound — All patients will undergo a cross-sectional imaging test as part of their standard of care at 3 and 6 months after surgery. A follow-up IUS will be performed within 18 months after index colonoscopy, as standard of care.
Diagnostic Test: Stool — Stool samples will be collected at 3 and 6 months after surgery and used for faecal calprotectin analysis. Research stool will be collected during the visit of index colonoscopy and at 12 months after index colonoscopy for metagenomics (only in Irish sites).
Diagnostic Test: Blood — Blood will be collected at 3 and 6 months after surgery and used as standard of care. Research blood will be collected during the visit of index colonoscopy and at 12 months after index colonoscopy for research - i.e. proteomic, genomic, cell experiments (only in Irish sites).
Diagnostic Test: Saliva — Saliva will be collected during the visit of index colonoscopy and at 12 months after surgery for research - i.e. optical spectroscopy (only in Irish site)
Other: Clinical follow-up — Patients will be followed-up at 6, 12 and 24 months after index endoscopy. Patients will be evaluated in clinic or by telephone call and the disease will be reassessed. The following scores will be repeated: Harvey Bradshaw Index (HBI) and CD Activity Index score (CDAI). Participants will give an update on their medication use.

SUMMARY:
This is a multicentre prospective international observational study. This study aims to introduce a novel multidimensional approach to precision imaging, enabling the identification and stratification of high-risk patients who can potentially benefit from early treatments to halt the progression of Crohn's disease (CD). The investigators will develop a novel endoscopic assessment system using endoscopic enhanced imaging (EEI) to evaluate early post-surgical changes and predict post-operative CD recurrence (POCr). By integrating with immune marker profiling, clinical data, and AI assessment of EEI and histology, the investigators further plan to improve risk stratification and reduce interobserver variability.

DETAILED DESCRIPTION:
Background:

Up to 70% of Crohn's disease (CD) patients will undergo a surgical resection in their lifetime. However, surgery is non-curative since 50% of patients have a recurrence, and about one-third need repeat surgery. The tools currently used to assess CD recurrences, such as faecal calprotectin (FCP), cross-sectional imaging (small bowel ultrasound, MRI scan) and conventional endoscopy, have a limited role in predicting early Post-Operative CD recurrence (POCr). Distinguishing inflammatory disease recurrence from post-surgical ischemic or suture-related alterations poses a significant challenge. Endoscopic Enhanced imaging (EEI) techniques like virtual electronic chromoendoscopy (VCE) and biopsy-like probe-based confocal laser endomicroscopy (pCLE) combined with artificial intelligence, can improve the detection of mucosal/vascular changes before major alterations become evident. VCE is available simply by switching a button. The pCLE probe will be passed through the endoscope channel like a biopsy forceps, enabling real-time, histology-like images of the intestine's lining and the gut barrier.

Study summary:

This is a multicentre prospective international observational study. This study aims to introduce a novel multidimensional approach to precision imaging, enabling the identification and stratification of high-risk patients who can potentially benefit from early treatments to halt the progression of CD.

The investigators will develop a novel endoscopic assessment system using EEI to evaluate early post-surgical changes and predict POCr. By integrating with immune marker profiling, clinical data, and AI assessment of EEI and histology, the investigators further plan to improve risk stratification and reduce interobserver variability. A detailed exploratory analysis will only be done in a cohort of patients in Ireland. The correlation between the new scoring system and established endoscopic and histologic scores, cross-sectional imaging, and non-invasive markers of inflammation will be evaluated. A multimodal machine learning model will be developed on EEI videos, histology, clinical data and immune molecular analysis to stratify patients' risk of early recurrence and long-term outcomes. The study will be divided into three phases:

* In the first phase, descriptor criteria for the assessment of post-operative Crohn's Disease will be defined. Gastroenterologists experienced in IBD endoscopy will review images and videos from an existing library showing the different grade of inflammation of the modified Rutgeerts score. These will be used for a stepwise discussion. A round table discussion using modified Delphi method will be conducted to ensure equal participation and identify the best component descriptors of endoscopic recurrence of CD. The components that achieved 100% consensus will be selected and the most important endoscopy predictive variables will be confirmed by using a machine learning technique. Finally, a new endoscopic score will be generated. Further, the investigators will first validate the new endoscopic score using the first 30 consecutive VCE and pCLE videos of POCr patients recruited in the multicenter PROSPER study. A structured consensus will be conducted with experts in Inflammatory Bowel Disease, endoscopy and histology to define the endoscopic findings of mucosal, vascular and intestinal barrier function. Subsequently, the investigators will prospectively validate the score in a large cohort of POCr patients enrolled in the PROSPER study and assess the diagnostic accuracy of the new scoring system in predicting post-surgical recurrence. Clinical information, blood, saliva, stool, and bowel specimens will be taken. Cross-sectional imaging (magnetic resonance imaging -MRI-, intestinal ultrasound -IUS-), endoscopy VCE and pCLE (in equipped centres) will be performed according to stool calprotectin 3 months after surgery. Patients will be followed up for 24 months and the results of the follow-up colonoscopy performed, as standard of care, within 18 months from the index colonoscopy, will be collected.
* In the second phase, the investigators will externally validate and reproduce the new scoring system by gastroenterologists using a computerized training module.
* In the third phase, an advanced computer-aided quantitative analysis of videos, images from VCE and pCLE, and digital histology will be developed and validated to enhance the prediction of POCr. Additionally, further machine learning models will be developed, utilizing comprehensive data from blood, stool, cross-sectional imaging, endoscopy, histology, immune markers, and OMICs to predict POCr and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 years and 75 years.
* Established diagnosis of CD at least six months prior to study.
* Patients who have undergone intestinal resection within 3 months before study entry or have surgery planned.

Exclusion Criteria:

* Inability to provide consent.
* Presence of serious co-morbidities (clinical contraindication).
* Presence of ostomy.
* Pregnancy or breastfeeding.
* Contraindication for colonoscopy or biopsies.
* Boston Bowel Preparation Scale Score <2 in the rectum plus left-sided colon.

Exclusion criteria for pCLE only:

* Allergy to nuts or shellfish.
* Severe or uncontrolled asthma.
* Use of beta blockers.
* Previous history of reaction to fluorescein.

Patients excluded from pCLE can still enter the study and undergo only standard-of-care endoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females aged between 18 and 75 years old and with an established diagnosis of CD, who have undergone surgery no more than three months before study entry, or have surgery planned, will be consecutively recruited after obtaining written consent. The sample size for the study is 225
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Early post-operative endoscopic recurrence | 3 months or 6 months
  Post surgical endoscopic recurrence will be defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) > 2 and Rutgeerts score > i2a
Early post-operative clinical recurrence | 3 months and 6 months
  Post surgical clinical recurrence will be defined as:
  * CD Activity Index score (CDAI) >200 and a >70-point increase from baseline, or
  * development of a new or re-draining fistula or abscess, or
  * requiring steroids, endoscopic dilatation, or hospitalization

SECONDARY OUTCOMES:
Post-operative clinical recurrence | 1 year and 2 years
  Post surgical clinical recurrence will be defined as:
  * CD Activity Index score (CDAI) >200 and a >70-point increase from baseline, or
  * development of a new or re-draining fistula or abscess, or
  * requiring steroids, endoscopic dilatation, or hospitalization and
  * new surgery at 12 and 24 months after colonoscopy.
Early post-operative histological recurrence | 3 months or 6 months
  Post surgical histologic recurrence will be defined as Robarts histopathology index (RHI) >3 and PICaSSO Histological remission Index (PHRI) > 0
Early post-operative IUS recurrence | 3 months or 6 months
  Post surgical IUS recurrence will be assessed according to:
  * Anastomotic bowel wall thickness (BWT)
  * Bowel wall stratification (BWS)
  * Lesion length
  * Presence of mesenteric lymphadenopathy
  * Proliferation of inflammatory mesenteric fat (iFat).
  * Presence of free fluid within the peritoneal cavity
  * Presence of strictures
  * Presence of fistulae
  * Presence of abscesses
  * Limberg score

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Iacucci, Professor, Study Chair — APC Microbiome Ireland, University College Cork
Locations (15):
- University of Leuven, Leuven, Belgium
- University of Calgary, Calgary, Canada
- University Hospital Erlangen, Erlangen, Germany
- Ireland (4):
  - Cork University Hospital, Cork
  - Mercy University Hospital, Cork
  - University College Dublin, Dublin
  - University College Hospitals Galway, Galway
- Rabin Medical Centre, Tel Aviv, Israel
- Italy (7):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - ASST Spedali Civili, Brescia
  - ASST Fatebenefratelli Sacco, Milan
  - IRCCS Cà Granda Ospedale Maggiore, Milan
  - University Vita-Salute San Raffaele, Milan
  - University Federico II, Naples
  - IRCCS San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349
- [Background] Gionchetti P, Dignass A, Danese S, Magro Dias FJ, Rogler G, Lakatos PL, Adamina M, Ardizzone S, Buskens CJ, Sebastian S, Laureti S, Sampietro GM, Vucelic B, van der Woude CJ, Barreiro-de Acosta M, Maaser C, Portela F, Vavricka SR, Gomollon F; ECCO. 3rd European Evidence-based Consensus on the Diagnosis and Management of Crohn's Disease 2016: Part 2: Surgical Management and Special Situations. J Crohns Colitis. 2017 Feb;11(2):135-149. doi: 10.1093/ecco-jcc/jjw169. Epub 2016 Sep 22. PMID 27660342
- [Background] Iacucci M, Ghosh S, Daperno M. Post-operative Recurrence of Crohn's Disease: There Is More to It than Meets the Eye. J Crohns Colitis. 2016 Sep;10(9):999-1000. doi: 10.1093/ecco-jcc/jjw094. Epub 2016 May 4. No abstract available. PMID 27147451
- [Background] Riviere P, Vermeire S, Irles-Depe M, Van Assche G, Rutgeerts P, de Buck van Overstraeten A, Denost Q, Wolthuis A, D'Hoore A, Laharie D, Ferrante M. No Change in Determining Crohn's Disease Recurrence or Need for Endoscopic or Surgical Intervention With Modification of the Rutgeerts' Scoring System. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1643-1645. doi: 10.1016/j.cgh.2018.09.047. Epub 2018 Oct 4. PMID 30291910
- [Background] Auzoux J, Boschetti G, Anon B, Aubourg A, Caulet M, Poisson L, Besson P, Lecomte T, Roger S, Picon L, Nancey S, Moussata D, Flourie B. Usefulness of confocal laser endomicroscopy for predicting postoperative recurrence in patients with Crohn's disease: a pilot study. Gastrointest Endosc. 2019 Jul;90(1):151-157. doi: 10.1016/j.gie.2019.02.030. Epub 2019 Mar 5. PMID 30849396
- [Background] Rispo A, Imperatore N, Testa A, Nardone OM, Luglio G, Caporaso N, Castiglione F. Diagnostic Accuracy of Ultrasonography in the Detection of Postsurgical Recurrence in Crohn's Disease: A Systematic Review with Meta-analysis. Inflamm Bowel Dis. 2018 Apr 23;24(5):977-988. doi: 10.1093/ibd/izy012. PMID 29688470
- [Background] Iacucci M, Cannatelli R, Parigi TL, Nardone OM, Tontini GE, Labarile N, Buda A, Rimondi A, Bazarova A, Bisschops R, Del Amor R, Meseguer P, Naranjo V, Ghosh S, Grisan E; PICaSSO group. A virtual chromoendoscopy artificial intelligence system to detect endoscopic and histologic activity/remission and predict clinical outcomes in ulcerative colitis. Endoscopy. 2023 Apr;55(4):332-341. doi: 10.1055/a-1960-3645. Epub 2022 Oct 13. PMID 36228649